CLINICAL TRIAL: NCT03417791
Title: Recovery of Serum Creatinine at Discharge Impacts Mortality, Long-term and Short-term
Brief Title: Recovery of Serum Creatinine at Discharge Impacts Mortality
Acronym: RECOST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GDREC2017296H
Record Dates: First submitted 2018-01-17; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2017-11

CONDITIONS: Kidney; Functional Disturbance
Keywords: recovery; serum creatinine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- kidney function recovery: the registry and follow up of consecutive patients with increased serum creatinine during hospital in 2007
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim of our study is to assess the mortality in the in-hospital patients who have elevated serum creatinine. A registry of patients with increased serum creatinine during hospital was conducted at the Guangdong General Hospital from January 1st, 2007 to December 30th, 2013. The primary clinical outcome is all-cause mortality, followed from the date of hospital discharge to Dec 30th 2018. Patients were divided into three groups, according to the serum creatinine recovery ratio (discharge/max serum creatinine). All-cause mortality, including the date of death, was identified from the electronic hospitalization data, phone follow-up, and confirmed by the household registration (HUKOU) system, a record of registration required by law in China. Baseline characteristics, including primary disease diagnosis, blood pressure, major treatment, drug use and et al, were collected. Demographic data were collected from the electronic hospitalization data and electronic hospital discharge records. All co-morbid conditions were identified using International Statistical Classification of Diseases, Tenth Revision (ICD-10), coding algorithms applied to electronic physician claims and electronic hospital discharge records.

ELIGIBILITY:
Inclusion Criteria:

* In-hospital patients in Guangdong General Hospital in 2007
* Age>=18y
* Patients with increased serum creatinine during hospital

Exclusion Criteria:

* Death during hospital
* Diagnosed with End-stage renal disease
* given the renal replace therapy during hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the registry and follow up of consecutive patients with increased serum creatinine during hospital in 2007
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 10 years
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Liming Yao, M.D., Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No